CLINICAL TRIAL: NCT00262704
Title: SimCare: Physician Intervention to Improve Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 0001600; R01HS010639 (AHRQ)
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Mellitus
Keywords: physician intervention; diabetes mellitus; primary care; quality improvement; disease management
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (No Intervention): Control group
- Group B (Active Comparator): Simulated case-based customized learning
  Interventions: Behavioral: Simulated case-based customized learning
- Group C (Active Comparator): Simulated case based customized learning + leader feedback
  Interventions: Behavioral: Simulated case based customized learning + leader feedback

INTERVENTIONS:
Behavioral: Simulated case-based customized learning — Formal Analysis of Diabetes Practice Style, Using SimCare cases with Process Trace Feedback
  Arms: Group B
Behavioral: Simulated case based customized learning + leader feedback — Formal Analysis of Diabetes Practice Style, Using SimCare cases with Process Trace Feedback + Physician Opinion Leader Feedback Tailored to Provider's Specific Practice Style
  Arms: Group C

SUMMARY:
This randomized trial will test the hypotheses that (a) a physician opinion leader intervention, (b) a "narrative process trace" physician feedback intervention, or (c) the combined intervention (a + b), are no more effective than (d) usual care in improving the clinical care of adult patients with type 2 diabetes.

DETAILED DESCRIPTION:
This randomized trial will test the hypothesis that (a) an influential physician feedback intervention, (b) a "narrative process trace" feedback intervention, or (c) the combined intervention (a + b), are no more effective than (d) usual care in improving the clinical care of adult patients with diabetes mellitus.

The unit of randomization and the unit of analysis will be primary care physicians who have more than 10 adult patients with diabetes mellitus. The 162 physicians eligible for this study provide care to about 6,804 adults with diagnosed diabetes at 24 primary care clinics. The narrative process trace intervention uses automated medical record (AMR)-mounted clinical cases to assess physicians' diabetes care decisions, with results provided as feedback to physicians. The influential physician feedback intervention emphasizes individualized education of physicians, which will be guided by the narrative process trace in the combined intervention group. Usual care includes the use of a diabetes clinical guideline, use of a diabetes patient registry that provides key clinical data for each adult patient with diabetes, and access to clinic-based diabetes education nurses. We have shown in previous controlled studies that the guideline, diabetes registry, and clinic-based diabetes education nurses have failed to significantly improve diabetes care on a population basis, thus justifying the additional, stronger interventions that now will be tested.

Dependent variables include glycemic control and cardiovascular risk reduction of all 3,360 patients cared for by the 80 study physicians. Secondary analysis will assess rates of screening for microvascular complications. Physicians will be randomized in blocks based on specialty, number of diabetes patients, and years of practice experience. Hierarchical data analysis will be used to accommodate the nested data and propensity scores will be used to correct for selection effects and missing data. Results of this experiment will advance our theoretical understanding of physician behavior change and quantify cost and impact of three specific intervention strategies to improve chronic disease care in the primary care setting. The study will have substantial impact on clinical practice and policy whether the results are positive or negative. If successful, the interventions will be easily disseminated to other primary care practice settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients- Diabetes patients associated with the n=57 physicians were selected according to the following criteria: (1) enrolled in HealthPartners on January 1, 1998, (2) be at least 19 years of age on January 1, 1998, (3) have an established diagnosis of diabetes mellitus in 1998 based on meeting at least one of the following two criteria: (a) have one or more inpatient, or two or more outpatient International Classification of Diseases-9 (ICD-9) diagnostic codes 250.xx for diabetes, or (b) have a filled prescription for a diabetes-specific drug including insulins, sulphonylureas, biguanides, alpha-glucosidase inhibitors, thiazolidinediones, or meglitinides.
* Physicians-All primary care adult care physicians (family physicians or primary care internists) employed full-time at HealthPartners medical groups as of 2000 were eligible for this study.

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2020 (Actual)
Dates: Start 2001-12; Primary Completion 2002-08 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
glycemic control | All A1c and LDL values and test dates were recorded for a defined 12-month period before and after the date of intervention for all diabetes patients under the care of study physicians
  Glycosylated hemoglobin (A1c) values and A1c test rates were used to assess glycemic control.
lipid control | All A1c and LDL values and test dates were recorded for a defined 12-month period before and after the date of intervention for all diabetes patients under the care of study physicians
  LDL-cholesterol levels and test rates were used to assess lipid control.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J O'Connor, MD MPH, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Research Foundation, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] O'Connor PJ, Sperl-Hillen JM, Johnson PE, Rush WA, Biltz G. Clinical Inertia and Outpatient Medical Errors. In: Henriksen K, Battles JB, Marks ES, Lewin DI, editors. Advances in Patient Safety: From Research to Implementation (Volume 2: Concepts and Methodology). Rockville (MD): Agency for Healthcare Research and Quality (US); 2005 Feb. Available from http://www.ncbi.nlm.nih.gov/books/NBK20513/ PMID 21249838
- [Background] Dutta P, Biltz GR, Johnson PE, Sperl-Hillen JM, Rush WA, Duncan JE, O'Connor PJ. SimCare: A Simulation Model to Investigate Physician Decision-Making in the Care of Patients with Type 2 Diabetes. In K. Henriksen, J. Battles, D. Lewin, and E. Marks. Advances in Patient Safety: From Research to Implementation. Rockville, MD. Agency for Healthcare Research and Quality (AHRQ). 2005; Vol.4: Programs, Tools, and Products; 179-192. <http://www.ahrq.gov/qual/advances/>
- [Background] O'Connor PJ, Sperl-Hillen JM, Johnson PE, Rush WA. Identification, Classification, and Frequency of Medical Errors in Outpatient Diabetes Care. In: Henriksen K, Battles JB, Marks ES, Lewin DI, editors. Advances in Patient Safety: From Research to Implementation (Volume 1: Research Findings). Rockville (MD): Agency for Healthcare Research and Quality (US); 2005 Feb. Available from http://www.ncbi.nlm.nih.gov/books/NBK20464/ PMID 21249801
- [Background] O'Connor PJ. Overcome clinical inertia to control systolic blood pressure. Arch Intern Med. 2003 Dec 8-22;163(22):2677-8. doi: 10.1001/archinte.163.22.2677. No abstract available. PMID 14662620
- [Background] O'Connor PJ. Setting evidence-based priorities for diabetes care improvement. Int J Qual Health Care. 2003 Aug;15(4):283-5. doi: 10.1093/intqhc/mzg062. No abstract available. PMID 12930043
- [Background] Johnson PE, Veazie PJ, Kochevar L, O'Connor PJ, Potthoff SJ, Verma D, Dutta P. Understanding variation in chronic disease outcomes. Health Care Manag Sci. 2002 Aug;5(3):175-89. doi: 10.1023/a:1019740401536. PMID 12363045
- [Background] O'Connor PJ. Patient archetypes, physician archetypes, and tailored diabetes care. J Am Board Fam Pract. 2002 Jul-Aug;15(4):334-7. No abstract available. PMID 12150470
- [Result] O'Connor PJ, Sperl-Hillen JM, Johnson PE, Rush WA, Asche SE, Dutta P, Biltz GR. Simulated physician learning intervention to improve safety and quality of diabetes care: a randomized trial. Diabetes Care. 2009 Apr;32(4):585-90. doi: 10.2337/dc08-0944. Epub 2009 Jan 26. PMID 19171723